CLINICAL TRIAL: NCT01629797
Title: Knowledge Evaluation and Assessment of the Effectiveness of an Education Intervention on Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Assistant Professor of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: STU64905
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acne Vulgaris (Other): Patients with Acne vulgaris will receive educational teaching on Acne
  Interventions: Behavioral: Educational script on Acne

INTERVENTIONS:
Behavioral: Educational script on Acne — An educational script on Acne will be presented by investigator

SUMMARY:
Acne vulgaris is a chronic inflammatory disorder of the skin in the pilosebaceous unit of the hair follicle, associated with oil production. It is found across skin types and is present in 85% of adolescents, representing a large affected population. Because of the universal nature of the disease, 36.3% of acne patients come from backgrounds other than Caucasian.

The purpose of this study is to examine patient knowledge about acne in different populations and to assess the effectiveness of a teaching intervention on acne knowledge. The investigators aim is to better understand and subsequently reduce any potential health disparities within the minority populations.

This project will evaluate differences in acne knowledge between different ethnic groups, and the efficacy of an educational intervention. Subjects will first complete a survey evaluating their knowledge of acne and how acne affects them psychosocially before an educational intervention. Immediately following the intervention, the patient's knowledge of acne will be evaluated again. Finally, two months after the intervention, a phone call will be made evaluating their retention of the education materials and their quality of life related to psychosocial effects of acne. Investigating this educational intervention and any current disparities in acne education and understanding will better allow us to educate and treat acne patients in the future.

ELIGIBILITY:
Inclusion criteria:

* Subjects ages 18 years of age and older and able to give consent
* Subjects with a diagnosis of acne vulgaris

Exclusion criteria:

* Subjects who are not proficient in English
* Subjects who were unable to give informed consent
* Subjects who do not have a diagnosis of acne vulgaris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Kundu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Callender VD. Acne in ethnic skin: special considerations for therapy. Dermatol Ther. 2004;17(2):184-95. doi: 10.1111/j.1396-0296.2004.04019.x. PMID 15113286
- [Background] Cheng CE, Irwin B, Mauriello D, Liang L, Pappert A, Kimball AB. Self-reported acne severity, treatment, and belief patterns across multiple racial and ethnic groups in adolescent students. Pediatr Dermatol. 2010 Sep-Oct;27(5):446-52. doi: 10.1111/j.1525-1470.2010.01286.x. Epub 2010 Aug 26. PMID 20796234
- [Background] Dreno B. Assessing quality of life in patients with acne vulgaris: implications for treatment. Am J Clin Dermatol. 2006;7(2):99-106. doi: 10.2165/00128071-200607020-00003. PMID 16605290
- [Background] Hanna S, Sharma J, Klotz J. Acne vulgaris: more than skin deep. Dermatol Online J. 2003 Aug;9(3):8. PMID 12952755
- [Background] Tan JK, Vasey K, Fung KY. Beliefs and perceptions of patients with acne. J Am Acad Dermatol. 2001 Mar;44(3):439-45. doi: 10.1067/mjd.2001.111340. PMID 11209112
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- See also: Northwestern University Department of Dermatology Actively Enrolling Research Trials — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Acne Vulgaris: Subjects completed a questionnaire assessing 26 items related to knowledge of acne pathogenesis, signs and symptoms of acne, risk factors for acne, and beliefs about acne. Next, subjects listened to a scripted, educational lecture about acne developed from the American Academy of Dermatology (AAD) acne educational materials. In addition, the AAD patient education pamphlet on acne was provided to each subject. Subjects completed the questionnaire to assess knowledge about acne immediately post-lecture. Two months after the educational lecture, subjects were contacted by phone to complete a final questionnaire to assess knowledge about acne.
Period: Overall Study
Arm/Group | Acne Vulgaris
Started | 100
Completed | 82
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Acne Vulgaris
Number analyzed (Participants) | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Correct Responses to Questionnaire Items Immediately Before and After and Educational Lecture
Description: In order to evaluate the immediate effect of an educational lecture about acne, subjects completed a questionnaire to assess knowledge about acne immediately before and after the educational lecture. The number of correct responses to each questionnaire item was calculated pre- and post-educational lecture.
Time Frame: immediately before and after an educational lecture
Measure: Number; unit: participants
Groups:
- Pre-educational Lecture; Post-educational Lecture: Subjects completed a questionnaire assessing 26 items related to knowledge of acne pathogenesis, signs and symptoms of acne, risk factors for acne, and beliefs about acne. Next, subjects listened to a scripted, educational lecture about acne developed from the American Academy of Dermatology (AAD) acne educational materials. In addition, the AAD patient education pamphlet on acne was provided to each subject. Subjects completed the questionnaire to assess knowledge about acne immediately post-lecture.
Arm/Group | Pre-educational Lecture | Post-educational Lecture
Number analyzed (Participants) | 100 | 100
participants
  How to wash skin | 79 | 79
  How often to wash face | 74 | 79
  Diet affects acne | 60 | 43
  Dirt affects acne | 31 | 37
  Hair product affects acne | 45 | 63
  Sweat affects acne | 27 | 43
  Cosmetics affect acne | 61 | 65
  Moisturizers affect acne | 40 | 43
  Humidity affects acne | 35 | 53
  Season affects acne | 44 | 63
  Stress affects acne | 72 | 76
  Drugs affect acne | 56 | 50
  Stress worsens acne | 72 | 76
  Diet worsens acne | 30 | 46
  Menses worsens acne | 64 | 77
  Hormones worsen acne | 68 | 76
  Genetics worsen acne | 48 | 66
  Excess oil causes acne | 67 | 77
  Clogged pores cause acne | 77 | 80
  Bacteria causes acne | 70 | 77
  Inflammation causes acne | 33 | 70
  Acne can be cured | 29 | 69
  Results of acne treatment | 38 | 70
  Acne treatment lasts | 45 | 61
  Acne can scar | 82 | 81
  Cosmetics worsen acne | 79 | 79

2. Secondary Outcome: Number of Correct Responses to Questionnaire Items Before and 2 Months After an Educational Lecture
Description: In order to evaluate the long-term effect of an educational lecture about acne, subjects completed a questionnaire to assess knowledge about acne immediately before and two months after the educational lecture. The number of correct responses to each questionnaire item was calculated pre- and two months post-educational lecture.
Time Frame: before and 2 months after an educational lecture
Measure: Number; unit: participants
Groups:
- Pre-educational Lecture; Two Months Post-educational Lecture: Subjects completed a questionnaire assessing 26 items related to knowledge of acne pathogenesis, signs and symptoms of acne, risk factors for acne, and beliefs about acne. Next, subjects listened to a scripted, educational lecture about acne developed from the American Academy of Dermatology (AAD) acne educational materials. In addition, the AAD patient education pamphlet on acne was provided to each subject. Subjects completed the questionnaire to assess knowledge about acne immediately post-lecture. Two months after the educational lecture, subjects were contacted by phone to complete a final questionnaire to assess knowledge about acne.
Arm/Group | Pre-educational Lecture | Two Months Post-educational Lecture
Number analyzed (Participants) | 100 | 82
participants
  How to wash skin | 79 | 78
  How often to wash face | 74 | 76
  Diet affects acne | 60 | 55
  Dirt affects acne | 31 | 12
  Hair product affects acne | 45 | 65
  Sweat affects acne | 27 | 22
  Cosmetics affect acne | 61 | 76
  Moisturizers affect acne | 40 | 58
  Humidity affects acne | 35 | 32
  Season affects acne | 44 | 36
  Stress affects acne | 77 | 77
  Drugs affect acne | 56 | 80
  Stress worsens acne | 72 | 77
  Diet worsens acne | 30 | 25
  Menses worsens acne | 64 | 76
  Hormones worsen acne | 68 | 79
  Genetics worsen acne | 48 | 63
  Excess oil causes acne | 67 | 81
  Clogged pores cause acne | 77 | 82
  Bacteria causes acne | 70 | 77
  Inflammation causes acne | 33 | 69
  Acne can be cured | 29 | 65
  Results of acne treatment | 38 | 47
  Acne treatment lasts | 45 | 43
  Acne can scar skin | 82 | 80
  Cosmetics worsen acne | 79 | 77

ADVERSE EVENTS:
Arm/Group | Acne Vulgaris
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes